CLINICAL TRIAL: NCT02323256
Title: Neurophysiological Measures During Sound and Speech Perception in Cochlear Implanted Patients and Development of New Speech Rehabilitation Tools
Brief Title: Neurophysiological Measures of Auditory Perception and Rehabilitation in Cochlear Implanted Patients
Acronym: NEUROSYLLABIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014.857; 2014-A00345-42 (Other: ANSM)
Record Dates: First submitted 2014-10-15; First posted 2014-12-23 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Deafness
Keywords: cochlear implant; deafness; audiometry; speech perception; severe to profound deafness restored with cochlear implantation
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- newly cochlear implanted adult patients (Experimental): longitudinal group
  Interventions: Other: Auditory steady-state response ASSR; Other: Speech-ABR; Other: Acoustic Change Complex ACC; Other: P1-N1-P2 complex and Mismatch Negativity MMN
- newly cochlear implanted children (Experimental): longitudinal group
  Interventions: Other: Auditory steady-state response ASSR; Other: Speech-ABR; Other: Acoustic Change Complex ACC; Other: P1-N1-P2 complex and Mismatch Negativity MMN
- cochlear implanted adult patients (CI>1 year) (Active Comparator): transversal group
  Interventions: Other: Auditory steady-state response ASSR; Other: Speech-ABR; Other: Acoustic Change Complex ACC; Other: P1-N1-P2 complex and Mismatch Negativity MMN
- normal hearing adult subjects (Active Comparator): transversal group
  Interventions: Other: Auditory steady-state response ASSR; Other: Speech-ABR; Other: Acoustic Change Complex ACC; Other: P1-N1-P2 complex and Mismatch Negativity MMN

INTERVENTIONS:
Other: Auditory steady-state response ASSR — comparison of ASSR amplitudes in response to amplitude-modulated sounds delivered at different intensities
Other: Speech-ABR
  Other Names: comparison of spectro-temporal analysis of speech-ABR generated in response to speech syllables
Other: Acoustic Change Complex ACC — comparison of ACC complex in response to changes within speech stimulation
Other: P1-N1-P2 complex and Mismatch Negativity MMN — comparison of amplitudes and latencies of P1-N1-P2 complex and MMN generated in response to the detection of changes in a series of auditory stimulation

SUMMARY:
This study aims at investigating new automatic fitting techniques for cochlear implant patients based on objective measures. For this reason, the evolution of these neurophysiological measures, expressing the encoding of pure tones and speech, will be characterized in cochlear implanted patients as a function of post-implantation time and will be compared to those of normal hearing subjects. Moreover, the effect of auditory training with new tools based on serious games will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* native French speaker
* no medical treatment for behavior or neurological disorders
* normal or corrected vision
* right-handed
* normal ORL examination
* valid affiliation to social security
* absence of participation to another study

For the cochlear implanted patients:

* aged from 1 to 70
* bilateral severe to profound deafness
* cochlear implant
* congenital deafness, pre or post lingual

For the normal-hearing subjects:

* Aged from 18 to 70
* Normal tonal audiometry

Exclusion Criteria:

* No signed consent
* Treatment for depression, epilepsy, Parkinson's or Alzheimer's disease
* Physical health deficiency
* Mental retardation
* Neurological or psychiatric disease incompatible with the testing procedure
* Schooling in a foreign language
* Foreign language spoken at home with both parents
* Invalid social security
* For the normal hearing subjects, no known hearing deficits

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Amplitude of auditory steady state responses ASSR | one year at least after CI activation
Spectro-temporal analysis of speech-ABR | one year at least after CI activation
Acoustic Change Complex ACC | one year at least after CI activation
  Amplitudes and latencies of ACC
amplitudes and latencies of P1/N1/P2 complex and Mismatch Negativity MMN | one year at least after CI activation
Evolution of amplitude of auditory steady state responses ASSR | 1 month, 3 months, 6 months, 9 months and 12 months after CI activation
  Evolution of ASSR amplitudes as a function of time during the first year of CI activation in newly implanted patients
Evolution of spectro-temporal analysis of speech-ABR | 1 month, 3 months, 6 months, 9 months and 12 months after CI activation
  Evolution of spectro-temporal analysis of speech-ABR as a function of time during the first year of CI activation in newly implanted patients
Acoustic Change Complex ACC | 1 month, 3 months, 6 months, 9 months and 12 months after CI activation
  Evolution of amplitudes and latencies of ACC as a function of time during the first year of CI activation in newly implanted patients
amplitudes and latencies of P1/N1/P2 complex and Mismatch Negativity MMN | 1 month, 3 months, 6 months, 9 months and 12 months after CI activation
  Evolution of amplitudes and latencies of P1N1P2 and MMN as a function of time during the first year of CI activation in newly implanted patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Attina V, Mina F, Stahl P, Duroc Y, Veuillet E, Truy E, Thai-Van H. A New Method to Test the Efficiency of Cochlear Implant Artifacts Removal From Auditory Evoked Potentials. IEEE Trans Neural Syst Rehabil Eng. 2017 Dec;25(12):2453-2460. doi: 10.1109/TNSRE.2017.2723952. Epub 2017 Jul 6. PMID 28692981